CLINICAL TRIAL: NCT00534469
Title: Autologous Bone Marrow Transplantation for Non-M3 Acute Myeloid Leukemia (AML) in First Remission in Patients </=60 Years of Age Using Busulfan/Fractionated Total Body Irradiation (FTBI) and VP16 as the Preparative Regimen
Brief Title: Auto BMT for Non-M3 AML in 1st Remission in Pts </=60y of Age Using Busulfan/FTBI & VP16 as a Prep R
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 99040; P30CA033572 (NIH); CHNMC-99040; CDR0000564772 (Registry Identifier: NCI PDQ)
Record Dates: First submitted 2007-09-20; First posted 2007-09-24 (Estimated); Results first posted 2023-03-21 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Leukemia
Keywords: adult acute myeloid leukemia in remission; adult acute myeloid leukemia with 11q23 (MLL) abnormalities; adult acute myeloid leukemia with inv(16)(p13;q22); adult acute myeloid leukemia with t(16;16)(p13;q22); adult acute myeloid leukemia with t(8;21)(q22;q22); adult acute basophilic leukemia; adult acute eosinophilic leukemia; adult erythroleukemia (M6a); adult pure erythroid leukemia (M6b); adult acute megakaryoblastic leukemia (M7); adult acute minimally differentiated myeloid leukemia (M0); adult acute monoblastic leukemia (M5a); adult acute monocytic leukemia (M5b); adult acute myeloblastic leukemia with maturation (M2); adult acute myeloblastic leukemia without maturation (M1); adult acute myelomonocytic leukemia (M4)
MeSH Terms: conditions — Leukemia; Congenital Abnormalities; Leukemia, Basophilic, Acute; Leukemia, Eosinophilic, Acute; Leukemia, Erythroblastic, Acute; Leukemia, Megakaryoblastic, Acute; Leukemia, Monocytic, Acute; Leukemia, Myeloid, Acute; Leukemia, Myelomonocytic, Acute | interventions — aldesleukin; Filgrastim; Busulfan; Cytarabine; Etoposide; Idarubicin; Bone Marrow Transplantation; Peripheral Blood Stem Cell Transplantation; Whole-Body Irradiation

ARMS (1):
- HD ARA-C with or without Idarubicin (Experimental): This study was designed as a single-arm study.
  Strata were:
  HD ARA-C w/ Idarubicin, CR<6 months N = 24 patients. HD ARA-C w/ Idarubicin, CR>6 months N=1. HD ARA-C consolidation, CR<6 months N=5. HD ARA-C consolidation, CR>6 months N= 0.
  Interventions: Biological: aldesleukin; Biological: filgrastim; Drug: busulfan; Drug: cytarabine; Drug: etoposide; Drug: idarubicin; Procedure: autologous hematopoietic stem cell transplantation; Procedure: bone marrow transplantation; Procedure: peripheral blood stem cell transplantation; Radiation: total-body irradiation

INTERVENTIONS:
Biological: aldesleukin
  Other Names: Proleukin
Biological: filgrastim
  Other Names: Neupogen
Drug: busulfan
  Other Names: Myleran; Busulfex IV
Drug: cytarabine
  Other Names: cytosine arabinoside; ara-C; arabinofuranosyl cytidine; Cytosar-U
Drug: etoposide
  Other Names: VP-16; Vepesid; Toposar; Etophosphos
Drug: idarubicin
  Other Names: Idamycin; Zavedos; 4-demethoxydaunorubicin
Procedure: autologous hematopoietic stem cell transplantation
Procedure: bone marrow transplantation
Procedure: peripheral blood stem cell transplantation
Radiation: total-body irradiation

SUMMARY:
RATIONALE: Giving chemotherapy before an autologous stem cell transplant stops the growth of cancer cells by stopping them from dividing or killing them. After treatment, stem cells are collected from the patient's blood and/or bone marrow and stored. More chemotherapy and radiation therapy is given to prepare the bone marrow for the stem cell transplant. The stem cells are then returned to the patient to replace the blood-forming cells that were destroyed by the chemotherapy and radiation therapy. Giving aldesleukin after transplant may help keep cancer cells from coming back after transplant.

PURPOSE: This phase II trial is studying the side effects and how well giving busulfan and etoposide together with total-body irradiation followed by autologous stem cell transplant and aldesleukin works in treating patients with acute myeloid leukemia in first remission.

DETAILED DESCRIPTION:
OBJECTIVES:

* To evaluate the efficacy and toxicity of a preparative regimen comprising busulfan, etoposide, and fractionated total-body irradiation followed by autologous stem cell transplantation and aldesleukin after treatment with consolidation therapy comprising high-dose cytarabine with or without idarubicin in patients with acute myeloid leukemia in first remission.
* To estimate the long-term disease-free survival of patients treated with this regimen.
* To further evaluate the effect of prognostic factors (e.g., cytogenetics, WBC at presentation, and number of courses of induction therapy required to achieve remission) on the outcome of autologous stem cell transplantation and targeted busulfan dose.

OUTLINE:

* Consolidation therapy: Patients who received prior consolidation therapy are evaluated to determine the need for additional consolidation therapy. Patients who have not received prior consolidation therapy receive high-dose cytarabine IV over 3 hours every 12 hours on days 1-4 and idarubicin* IV over 5-10 minutes on days 1-3.

NOTE: *Patients with good risk cytogenetics t(8;21), inv(16), or t(16;16) or patients who received > 200 mg/m² of anthracycline do not receive idarubicin.

* Stem cell collection: All patients receive filgrastim (G-CSF) IV or subcutaneously (SC) twice daily beginning 7 days after completion of high-dose cytarabine and continuing until peripheral blood stem cell (PBSC) collection is completed. Patients who do not have an adequate number of PBSCs collected also undergo bone marrow collection.
* Preparative regimen: Patients receive busulfan IV over 2 hours on days -13 and -11 to -7 and etoposide IV on day -2. Patients also undergo fractionated total-body irradiation on days -6 to -3 for a total of 8-10 fractions.
* Autologous stem cell transplantation: Patients undergo autologous stem cell transplantation using PBSCs (with or without bone marrow) on day 0. Patients receive G-CSF IV or SC daily beginning on day 5 and continuing until blood counts recover.
* Interleukin therapy: Within 100 days post-transplantation, patients receive aldesleukin IV continuously on days 1-4 and 9-18.

After completion of study treatment, patients are followed periodically.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of acute myeloid leukemia (AML)

  * FAB types M0-2 and M4-M7

    * No M3 disease
* In first complete hematological remission as confirmed by marrow aspiration and biopsy

  * No cytogenetic abnormality in the remission marrow
  * In complete remission for less than 6 months

    * Patients who have been in complete remission for more than 6 months may be eligible upon approval of the principal investigator
* No prior myeloproliferative disorder (e.g., chronic myeloid leukemia, myelofibrosis, essential thrombocytosis, or polycythemia vera)
* No prior myelodysplasia or secondary leukemia

PATIENT CHARACTERISTICS:

* FEV_1 > 60%
* DLCO > 50%
* Cardiac ejection fraction ≥ 50%
* Creatinine clearance > 60 mL/min
* No severe chronic medical or psychological illness that, in the judgement of the principal investigator, would jeopardize the ability of the patient to tolerate aggressive chemotherapy
* No HIV positivity
* Not pregnant
* Negative pregnancy test

PRIOR CONCURRENT THERAPY:

* Prior consolidation therapy allowed
* No concurrent use the following medications during aldesleukin therapy :

  * Corticosteroids (including blood product "pre-meds")
  * Pentoxifylline
  * IV or intrathecal methotrexate
  * IV immunoglobulin
  * Other cytokines or growth factors

Ages: 16 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Actual)
Dates: Start 2000-02-08 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2025-07-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anthony S. Stein, MD, Study Chair — City of Hope Comprehensive Cancer Center

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 60 patients went on-study. 52 went on to autologous transplant. Seven completed consolidation therapy without moving on to transplant. One was given an allogeneic transplant.
Groups:
- HD ARA-C With Idarubicin, or Without Idarubicin if Previously Treated With an Anthracycline.: HD ARA-C with Idarubicin Consolidation, Busulfan/FTBI/VP16/PSC/BMT
  aldesleukin
  filgrastim
  busulfan
  cytarabine
  etoposide
  idarubicin
  autologous hematopoietic stem cell transplantation
  peripheral blood stem cell transplantation
  total-body irradiation
Period: Overall Study
Arm/Group | HD ARA-C With Idarubicin, or Without Idarubicin if Previously Treated With an Anthracycline.
Started | 52
Completed | 52
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Patients who went on to autologous transplant.
Arm/Group | HD ARA-C With Idarubicin, or Without Idarubicin if Previously Treated With an Anthracycline.
Number analyzed (Participants) | 52
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 2
  Between 18 and 65 years | 50
  >=65 years | 0
Age, Continuous [Median (Full Range); unit: years] | 42.3 [16.5 to 59.7]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31
  Male | 21
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/Ethnicity: American Indian or Alaska Native, not of Hispanic Origin | 1
  Race/Ethnicity: Asian or Pacific Islander, not of Hispanic Origin | 3
  Race/Ethnicity: Black, not of Hispanic Origin | 2
  Race/Ethnicity: Hispanic | 6
  Race/Ethnicity: White, not of Hispanic Origin | 40
Region of Enrollment [Number; unit: participants] — Country of enrollment: USA
  participants
    United States | 52

OUTCOME MEASURES:

1. Primary Outcome: Disease-Free Survival at 2-Year Post-Transplant
Description: Kaplan-Meier estimates at 2-years post-transplant, with 95% confidence intervals based on logit limit transformation of Greenwood's variance. Outcome is death or relapse, censor is alive in continual complete remission at the date of last clinical disease assessment.
Time Frame: Estimate at 2 years post treatment
Population: Transplanted patients
Measure: Number (95% Confidence Interval); unit: Proportion of pts alive in remission
Groups:
- HD ARA-C Intermediate Cytogenetics: HD ARA-C Consolidation, Busulfan/FTBI/VP16/PSC/BMT +/- Idarubicin
  aldesleukin
  filgrastim
  busulfan
  cytarabine
  etoposide
  idarubicin
  autologous hematopoietic stem cell transplantation
  bone marrow transplantation
  peripheral blood stem cell transplantation
  total-body irradiation
Arm/Group | HD ARA-C Intermediate Cytogenetics
Number analyzed (Participants) | 52
Proportion of pts alive in remission | 0.65 [0.52 to 0.77]

2. Secondary Outcome: Disease-Free Survival at 2-Year Post-Transplant by Cytogenetic Risk
Description: as for outcome 1
Time Frame: Kaplan-Meier estimate 2 years post treatment
Measure: Number (95% Confidence Interval); unit: Proportion of pts alive in remission
Groups:
- Unfavorable Risk Cytogenetics; Intermediate Risk Cytogenetics; Favorable Risk Cytogenetics; Unknown Risk: Rejected Cytogenetics Study: Cytogenetic risk was estimated using criteria in effect in 1999.
Arm/Group | Unfavorable Risk Cytogenetics | Intermediate Risk Cytogenetics | Favorable Risk Cytogenetics | Unknown Risk: Rejected Cytogenetics Study
Number analyzed (Participants) | 3 | 20 | 11 | 6
Proportion of pts alive in remission | 0.33 [0.04 to 0.85] | 0.75 [0.52 to 0.89] | 0.75 [0.44 to 0.92] | 0.73 [0.41 to 0.91]
Statistical Analysis 1: Comparison: Unfavorable Risk Cytogenetics vs Intermediate Risk Cytogenetics vs Favorable Risk Cytogenetics vs Unknown Risk: Rejected Cytogenetics Study; Null hypothesis: All four groups are drawn from the same distribution. Alternative hypothesis: At least one of the groups has measurably different survival from the others; Test type: Other — Two-sided test; p = 0.43, Log Rank — Log-rank test (Mantel-Haenszel test). This p-value is not adjusted for multiple comparisons. The a priori threshold for statistical significance is 0.05

ADVERSE EVENTS:
Time Frame: Adverse Events monitored/assessed up to 1 year post-transplant. All-Cause Mortality monitored/assessed up to 19 years post-transplant.
Groups:
- HD ARA-C With or Without Idarubicin: This study was designed as a single-arm study.
  Strata were:
  HD ARA-C w/ Idarubicin, CR<6 months N = 24 patients. HD ARA-C w/ Idarubicin, CR>6 months N=1. HD ARA-C consolidation, CR<6 months N=5. HD ARA-C consolidation, CR>6 months N= 0.
  aldesleukin
  filgrastim
  busulfan
  cytarabine
  etoposide
  idarubicin
  autologous hematopoietic stem cell transplantation
  bone marrow transplantation
  peripheral blood stem cell transplantation
  total-body irradiation
Arm/Group | HD ARA-C With or Without Idarubicin
All-Cause Mortality (participants affected / at risk) | 37/60
Serious Adverse Events (participants affected / at risk) | 6/60
Other Adverse Events (participants affected / at risk) | 47/60
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | HD ARA-C With or Without Idarubicin (N=60)
Cardiac General - Other: CARDIOGENIC SHOCK (Cardiac disorders) | 1
Cardiac General - Other: CONGESTIVE HEART FAILURE (Cardiac disorders) | 1
Cardiac ischemia/infarction (Cardiac disorders) | 1
Myocarditis (Cardiac disorders) | 1
Febrile neutropenia (fever of unknown origin) (Infections and infestations) | 1
Infection, Bacterial (COH) (Infections and infestations) | 1
Adult Respiratory Distress Syndrome (ARDS) (Respiratory, thoracic and mediastinal disorders) | 2
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary/Upper Respiratory - Other: PULMONARY HYPERTENSION (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary/Upper Respiratory - Other: RESPIRATORY FAILURE DUE TO PULMONARY FIBROSIS (Respiratory, thoracic and mediastinal disorders) | 1
Renal/Genitourinary - Other: HEMORRHAGIC CYSTITIS (Renal and urinary disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | HD ARA-C With or Without Idarubicin (N=60)
Allergic reaction/hypersensitivity (including drug fever) (Immune system disorders) | 4
Allergic rhinitis (including sneezing, nasal stuffiness, postnasal drip) (Immune system disorders) | 2
Allergy/Immunology - Other: CHILLS AFTER I.V. AMPHOTERICIN INFUSION (Immune system disorders) | 1
Allergy/Immunology - Other: NASAL CONGESTION (Immune system disorders) | 1
Auditory/Ear - Other: DECREASED HEARING (Ear and labyrinth disorders) | 2
Auditory/Ear - Other: DECREASED HEARING AT RT. EAR (Ear and labyrinth disorders) | 1
Auditory/Ear - Other: MILD SENSORY NERVE LOSS AT HEARING (Ear and labyrinth disorders) | 1
Auditory/Ear - Other: RT. TYMPANIC MEMBRANE DULLNESS (Ear and labyrinth disorders) | 1
Veno-Occlusive Disease (VOD) (General disorders) | 1
Blood/Bone Marrow - Other: (Blood and lymphatic system disorders) | 1
Blood/Bone Marrow - Other: CHILLS UPON PRBC TRANSFUSION (Blood and lymphatic system disorders) | 1
Blood/Bone Marrow - Other: ENGRAFTMENT SYNDROME (Blood and lymphatic system disorders) | 1
Blood/Bone Marrow - Other: INCREASED MCV (Blood and lymphatic system disorders) | 1
Blood/Bone Marrow - Other: SPHEROCYTOSIS (Blood and lymphatic system disorders) | 1
Blood/Bone Marrow - Other: TRANSFUSION REACTION (Blood and lymphatic system disorders) | 1
Bone marrow cellularity (Blood and lymphatic system disorders) | 1
Hemoglobin (Blood and lymphatic system disorders) | 41
Leukocytes (total WBC) for BMT studies, if specified in the protocol. (Blood and lymphatic system disorders) | 46
Lymphopenia (Blood and lymphatic system disorders) | 35
Neutrophils/granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 1
Neutrophils/granulocytes (ANC/AGC) for BMT studies, if specified in the protocol. (Blood and lymphatic system disorders) | 45
Platelets (Blood and lymphatic system disorders) | 1
Platelets for BMT studies, if specified in the protocol. (Blood and lymphatic system disorders) | 43
Transfusion: Platelets for BMT studies, if specified in the protocol. (Blood and lymphatic system disorders) | 43
Transfusion: pRBCs (Blood and lymphatic system disorders) | 1
Transfusion: pRBCs for BMT studies, if specified in the protocol. (Blood and lymphatic system disorders) | 43
Cardiac Arrhythmia - Other: (Cardiac disorders) | 1
Cardiac Arrhythmia - Other: SOFT SYSTOLIC MURMUR GRADE 1/6 (Cardiac disorders) | 1
Palpitations (Cardiac disorders) | 2
Prolonged QTc interval (Cardiac disorders) | 1
Supraventricular and nodal arrhythmia (Cardiac disorders) | 27
Vasovagal episode (Cardiac disorders) | 1
Cardiac General - Other: ASCITES (Cardiac disorders) | 1
Cardiac General - Other: CARDIOMEGALY (Cardiac disorders) | 2
Cardiac General - Other: CHEST WALL SWELLING (Cardiac disorders) | 1
Cardiac General - Other: FACIAL EDEMA (Cardiac disorders) | 1
Cardiac General - Other: JUGULAR VENOUS DISTENSION INCREASED (Cardiac disorders) | 1
Cardiac General - Other: PERIORBITAL EDEMA (Cardiac disorders) | 1
Cardiac General - Other: RIGHT VENTRICULAR ENLARGEMENT (Cardiac disorders) | 1
Cardiac troponin I (cTnI) (Cardiac disorders) | 1
Hypertension (Cardiac disorders) | 8
Hypotension (Cardiac disorders) | 25
Left ventricular systolic dysfunction (Cardiac disorders) | 1
Pericardial effusion (non-malignant) (Cardiac disorders) | 3
Edema (Vascular disorders) | 23
INR (International Normalized Ratio of prothrombin time) (Blood and lymphatic system disorders) | 3
PTT (Partial Thromboplastin Time) (Blood and lymphatic system disorders) | 1
Constitutional Symptoms - Other: CHILLS (General disorders) | 1
Constitutional Symptoms - Other: FEVER (ABSENT NEUTROPENIA) (General disorders) | 1
Constitutional Symptoms - Other: VAGINAL ITCHINESS (General disorders) | 1
Fatigue (asthenia, lethargy, malaise) (General disorders) | 39
Fever (in the absence of neutropenia, where neutropenia is defined as ANC <1.0 x 10e9/L) (General disorders) | 29
Insomnia (General disorders) | 24
Rigors/chills (General disorders) | 30
Sweating (diaphoresis) (General disorders) | 2
Weight gain (General disorders) | 6
Weight loss (General disorders) | 27
Bruising (in absence of Grade 3 or 4 thrombocytopenia) (Skin and subcutaneous tissue disorders) | 1
Dermatology/Skin - Other: ABRASIONS ON KNUCKLES (Skin and subcutaneous tissue disorders) | 1
Dermatology/Skin - Other: BLISTERS ON THE TONGUE (Skin and subcutaneous tissue disorders) | 1
Dermatology/Skin - Other: BURN ON THIGH (FROM A SOUP) (Skin and subcutaneous tissue disorders) | 1
Dermatology/Skin - Other: BURNING FROM RADIATION (Skin and subcutaneous tissue disorders) | 1
Dermatology/Skin - Other: CRUST AT HICKMAN EXIT SITE (Skin and subcutaneous tissue disorders) | 1
Dermatology/Skin - Other: DECUBITUS ULCER (Skin and subcutaneous tissue disorders) | 1
Dermatology/Skin - Other: DERMATITIS FOCAL (Skin and subcutaneous tissue disorders) | 2
Dermatology/Skin - Other: DERMATITIS FOCAL (FINGER) (Skin and subcutaneous tissue disorders) | 1
Dermatology/Skin - Other: DRY LIPS (Skin and subcutaneous tissue disorders) | 1
Dermatology/Skin - Other: DRY SKIN (Skin and subcutaneous tissue disorders) | 1
Dermatology/Skin - Other: ERYTHEMA AT HICKMAN CATHETER EXIT SITE (Skin and subcutaneous tissue disorders) | 1
Dermatology/Skin - Other: ERYTHEMA AT HICKMAN EXIT SITE (Skin and subcutaneous tissue disorders) | 1
Dermatology/Skin - Other: ERYTHEMATOUS PALMS (Skin and subcutaneous tissue disorders) | 1
Dermatology/Skin - Other: EYELID SWELLING (Skin and subcutaneous tissue disorders) | 1
Dermatology/Skin - Other: FACIAL ERYTHEMA (Skin and subcutaneous tissue disorders) | 1
Dermatology/Skin - Other: HANDS SKIN REACTION (Skin and subcutaneous tissue disorders) | 1
Dermatology/Skin - Other: HICKMAN SITE TENDERNESS (Skin and subcutaneous tissue disorders) | 1
Dermatology/Skin - Other: HYPERPIGMENTED SKIN (Skin and subcutaneous tissue disorders) | 1
Dermatology/Skin - Other: IRRITATION AT HICKMAN EXIT SITE (Skin and subcutaneous tissue disorders) | 1
Dermatology/Skin - Other: IRRITATION OF SKIN FROM HICKMAN CATHETER TAPE (Skin and subcutaneous tissue disorders) | 1
Dermatology/Skin - Other: IRRITATION OF THE SKIN ALONG THE HICKMAN CATHETER SITE (Skin and subcutaneous tissue disorders) | 1
Dermatology/Skin - Other: LESION ON THE EYE CORNER (Skin and subcutaneous tissue disorders) | 1
Dermatology/Skin - Other: LESION ON UPPER LIP (HERPES) (Skin and subcutaneous tissue disorders) | 1
Dermatology/Skin - Other: LESIONS ON LIPS-HERPETIC (Skin and subcutaneous tissue disorders) | 1
Dermatology/Skin - Other: LICHENOID CHANGES OVER THE BUCCAL MUCOSA (Skin and subcutaneous tissue disorders) | 1
Dermatology/Skin - Other: LT. KNEE CONTRACTURE (Skin and subcutaneous tissue disorders) | 1
Dermatology/Skin - Other: NASAL CELLULITIS (Skin and subcutaneous tissue disorders) | 1
Dermatology/Skin - Other: PALE SKIN (Skin and subcutaneous tissue disorders) | 1
Dermatology/Skin - Other: PALLOR (PALE SKIN) (Skin and subcutaneous tissue disorders) | 1
Dermatology/Skin - Other: PALMAR ERYTHEMA (Skin and subcutaneous tissue disorders) | 1
Dermatology/Skin - Other: PEELING NAILS (Skin and subcutaneous tissue disorders) | 1
Dermatology/Skin - Other: PRURITUS UPON PLATELETS TRANSFUSION (Skin and subcutaneous tissue disorders) | 1
Dermatology/Skin - Other: RASH OVER THE GROIN AREA (Skin and subcutaneous tissue disorders) | 1
Dermatology/Skin - Other: RAW RECTAL AREA (Skin and subcutaneous tissue disorders) | 1
Dermatology/Skin - Other: REDDENED 2ND LT. TOE DUE TO OVERCLIPPING (Skin and subcutaneous tissue disorders) | 1
Dermatology/Skin - Other: REDDENED RAC EXIT SITE (Skin and subcutaneous tissue disorders) | 1
Dermatology/Skin - Other: REDNESS AT HICKMAN CATHETER EXIT SITE (Skin and subcutaneous tissue disorders) | 2
Dermatology/Skin - Other: REDNESS AT HICKMAN CATHETER SITE (Skin and subcutaneous tissue disorders) | 1
Dermatology/Skin - Other: REDNESS OF SKIN AT HICKMAN CATHETER SITE (Skin and subcutaneous tissue disorders) | 1
Dermatology/Skin - Other: REDNESS OF THE SKIN AT HICKMAN CATHETER SITE (Skin and subcutaneous tissue disorders) | 1
Dermatology/Skin - Other: SCROTAL AREA EXCORIATION (Skin and subcutaneous tissue disorders) | 1
Dermatology/Skin - Other: SCROTAL AREA PAIN (Skin and subcutaneous tissue disorders) | 1
Dermatology/Skin - Other: SCROTAL EXCORIATION (Skin and subcutaneous tissue disorders) | 1
Dermatology/Skin - Other: SHOULDER PAIN (Skin and subcutaneous tissue disorders) | 1
Dermatology/Skin - Other: SKIN CHANGES (Skin and subcutaneous tissue disorders) | 1
Dermatology/Skin - Other: SKIN EXCORIATION (Skin and subcutaneous tissue disorders) | 1
Dermatology/Skin - Other: SKIN INDURATION (PALMS) (Skin and subcutaneous tissue disorders) | 1
Dermatology/Skin - Other: SKIN LESION (Skin and subcutaneous tissue disorders) | 1
Dermatology/Skin - Other: SKIN LESIONS (Skin and subcutaneous tissue disorders) | 1
Dermatology/Skin - Other: SLIGHT SKIN EROSION DUE TO TAPE (Skin and subcutaneous tissue disorders) | 1
Dermatology/Skin - Other: SMALL CYST IN AXILLA (Skin and subcutaneous tissue disorders) | 1
Dermatology/Skin - Other: SWELLING AT CATHETER PORT (Skin and subcutaneous tissue disorders) | 1
Dermatology/Skin - Other: SWOLLEN RAC EXIT SITE (Skin and subcutaneous tissue disorders) | 1
Dermatology/Skin - Other: TENDERNESS ON SOLES AND PALMS (Skin and subcutaneous tissue disorders) | 1
Dermatology/Skin - Other: VAD SITE LEAKAGE (Skin and subcutaneous tissue disorders) | 1
Dermatology/Skin - Other: VITILIGO (Skin and subcutaneous tissue disorders) | 1
Dermatology/Skin - Other: WARM AND RED SKIN (Skin and subcutaneous tissue disorders) | 1
Dermatology/Skin - Other: WARM SKIN (Skin and subcutaneous tissue disorders) | 1
Dermatology/Skin - Other: YELLOWISH DRAINAGE FROM RAC EXIT SITE (Skin and subcutaneous tissue disorders) | 1
Dry skin (Skin and subcutaneous tissue disorders) | 23
Flushing (Skin and subcutaneous tissue disorders) | 15
Hair loss/alopecia (scalp or body) (Skin and subcutaneous tissue disorders) | 12
Injection site reaction/extravasation changes (Skin and subcutaneous tissue disorders) | 10
Nail changes (Skin and subcutaneous tissue disorders) | 1
Pigmentation changes (e.g., vitiligo) (Skin and subcutaneous tissue disorders) | 10
Pruritus/itching (Skin and subcutaneous tissue disorders) | 22
Rash/dermatitis associated with high-dose chemotherapy or BMT studies. (Skin and subcutaneous tissue disorders) | 3
Rash/desquamation (Skin and subcutaneous tissue disorders) | 14
Rash/desquamation associated with graft versus host disease (GVHD) (Skin and subcutaneous tissue disorders) | 22
Rash: hand-foot skin reaction (Skin and subcutaneous tissue disorders) | 12
Hot flashes/flushes (Endocrine disorders) | 1
Anorexia (Gastrointestinal disorders) | 40
Ascites (non-malignant) (Gastrointestinal disorders) | 1
Colitis (Gastrointestinal disorders) | 2
Constipation (Gastrointestinal disorders) | 4
Dehydration (Gastrointestinal disorders) | 8
Diarrhea (Gastrointestinal disorders) | 19
Diarrhea associated with graft versus host disease (GVHD) (Gastrointestinal disorders) | 20
Dry mouth/salivary gland (xerostomia) (Gastrointestinal disorders) | 13
Dysphagia-esophageal related to radiation (Gastrointestinal disorders) | 2
Esophagitis (Gastrointestinal disorders) | 30
Flatulence (Gastrointestinal disorders) | 3
Gastritis (including bile reflux gastritis) (Gastrointestinal disorders) | 2
Gastrointestinal - Other: ABD. BLOATING (Gastrointestinal disorders) | 1
Gastrointestinal - Other: ABDOMINAL BLOATING (Gastrointestinal disorders) | 1
Gastrointestinal - Other: ABDOMINAL DISTENTION (Gastrointestinal disorders) | 1
Gastrointestinal - Other: BLOATING (Gastrointestinal disorders) | 2
Gastrointestinal - Other: DECREASED GASTRIC EMPTYING (Gastrointestinal disorders) | 1
Gastrointestinal - Other: DELAYED GASTRIC EMPTYING (Gastrointestinal disorders) | 1
Gastrointestinal - Other: DIARRHEA (Gastrointestinal disorders) | 1
Gastrointestinal - Other: DIARRHEA FOR BMT (Gastrointestinal disorders) | 1
Gastrointestinal - Other: DRY HEAVES (Gastrointestinal disorders) | 2
Gastrointestinal - Other: ESOPHAGITIS (Gastrointestinal disorders) | 1
Gastrointestinal - Other: FULLNESS IN RUQ (Gastrointestinal disorders) | 1
Gastrointestinal - Other: GAGGING (Gastrointestinal disorders) | 1
Gastrointestinal - Other: GALL BLADDER SLUDGE (US) (Gastrointestinal disorders) | 1
Gastrointestinal - Other: HEMORRHOID (Gastrointestinal disorders) | 2
Gastrointestinal - Other: HEPATOMEGALY (Gastrointestinal disorders) | 1
Gastrointestinal - Other: INCREASED MOUTH SECRETION (Gastrointestinal disorders) | 1
Gastrointestinal - Other: INCREASED MUCUS SECRETION (Gastrointestinal disorders) | 1
Gastrointestinal - Other: INCREASED ORAL MUCOUS SECRETION (Gastrointestinal disorders) | 1
Gastrointestinal - Other: INCREASED PHARYNGEAL SECRETION (Gastrointestinal disorders) | 1
Gastrointestinal - Other: INCREASED SALIVARY SECRETION (Gastrointestinal disorders) | 1
Gastrointestinal - Other: INCREASED SALIVATION (Gastrointestinal disorders) | 2
Gastrointestinal - Other: INCREASED SECRETION OF MOUTH AND PHARYNX (Gastrointestinal disorders) | 1
Gastrointestinal - Other: INDIGESTION (Gastrointestinal disorders) | 2
Gastrointestinal - Other: IRRITATION ALONG THE SIDES OF TONGUE (Gastrointestinal disorders) | 1
Gastrointestinal - Other: IRRITATION OF THROAT (Gastrointestinal disorders) | 1
Gastrointestinal - Other: ITCHINESS OF THROAT (Gastrointestinal disorders) | 1
Gastrointestinal - Other: LEFT CHEECK SWELLING (Gastrointestinal disorders) | 1
Gastrointestinal - Other: MUCOSITIS TONGUE (Gastrointestinal disorders) | 5
Gastrointestinal - Other: ORAL THRUSH (Gastrointestinal disorders) | 1
Gastrointestinal - Other: RETCHING (Gastrointestinal disorders) | 1
Gastrointestinal - Other: SLIGHT BULGE OF ABDOMEN DUE TO VALSALVA MANEUVER (Gastrointestinal disorders) | 1
Gastrointestinal - Other: SLIGHT HYPERTHROPHY OF TONGUE PAPILLAE (Gastrointestinal disorders) | 1
Gastrointestinal - Other: SLIGHT YELLOW CLOUDING ON TONGUE (Gastrointestinal disorders) | 1
Gastrointestinal - Other: SLOUGHING OF ORAL BUCCAL MUCOSA (Gastrointestinal disorders) | 1
Gastrointestinal - Other: SLOUGHING OF THICK WHITE FILM FROM TONGUE (Gastrointestinal disorders) | 1
Gastrointestinal - Other: SLOUGHING OF TONGUE MUCOSA (Gastrointestinal disorders) | 1
Gastrointestinal - Other: SPLENOMEGALY (Gastrointestinal disorders) | 1
Gastrointestinal - Other: STOMACH DISCOMFORT (Gastrointestinal disorders) | 1
Gastrointestinal - Other: SUBMANDIBULAR AREA SWELLING (Gastrointestinal disorders) | 1
Gastrointestinal - Other: SUPERFICIAL ULCERATION OF BOTH TONSILS (Gastrointestinal disorders) | 1
Gastrointestinal - Other: SWOLLEN TONGUE (Gastrointestinal disorders) | 1
Gastrointestinal - Other: TENDERNESS OF LOWER ABDOMEN (Gastrointestinal disorders) | 1
Gastrointestinal - Other: THIRSTY (Gastrointestinal disorders) | 1
Gastrointestinal - Other: THROAT CONGESTION (Gastrointestinal disorders) | 1
Gastrointestinal - Other: TONGUE MUCOSITIS (Gastrointestinal disorders) | 2
Gastrointestinal - Other: UNABLE TO SWALLOW MOUTH SECRETION (Gastrointestinal disorders) | 1
Gastrointestinal - Other: UNABLE TO SWALLOW SECRETION (Gastrointestinal disorders) | 1
Gastrointestinal - Other: VOMITING OF BLOODY MUCUS AND TISSUE (Gastrointestinal disorders) | 1
Heartburn/dyspepsia (Gastrointestinal disorders) | 25
Ileus, GI (functional obstruction of bowel, i.e., neuroconstipation) (Gastrointestinal disorders) | 2
Mucositis/stomatitis (functional/symptomatic) (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 43
Proctitis (Gastrointestinal disorders) | 1
Salivary gland changes/saliva (Gastrointestinal disorders) | 15
Stomatitis/pharyngitis (oral/pharyngeal mucositis) (Gastrointestinal disorders) | 41
Taste alteration (dysgeusia) (Gastrointestinal disorders) | 8
Vomiting (Gastrointestinal disorders) | 42
Hematemesis (Vascular disorders) | 12
Hematuria (in the absence of vaginal bleeding) (Vascular disorders) | 8
Hemoptysis (Vascular disorders) | 5
Hemorrhage/bleeding with grade 3 or 4 thrombocytopenia (Vascular disorders) | 23
Hemorrhage/bleeding without grade 3 or 4 thrombocytopenia (Vascular disorders) | 13
Melena/GI bleeding (Vascular disorders) | 4
Rectal bleeding/hematochezia (Vascular disorders) | 4
Hemorrhage, GU (Vascular disorders) | 13
Hemorrhage, pulmonary/upper respiratory (Vascular disorders) | 22
Hemorrhage/Bleeding - Other: BLEEDING FROM DECUBITUS AREA (Vascular disorders) | 1
Hemorrhage/Bleeding - Other: BLEEDING FROM HICKMAN CATHETER SITE (Vascular disorders) | 1
Hemorrhage/Bleeding - Other: BLEEDING FROM MOUTH (Vascular disorders) | 1
Hemorrhage/Bleeding - Other: BLEEDING FROM PHARYNX (Vascular disorders) | 1
Hemorrhage/Bleeding - Other: BLEEDING FROM RAC SITE (Vascular disorders) | 1
Hemorrhage/Bleeding - Other: BLEEDING FROM THE SKIN (SCATCH) (Vascular disorders) | 1
Hemorrhage/Bleeding - Other: BLEEDING FROM THROAT (Vascular disorders) | 1
Hemorrhage/Bleeding - Other: BLEEDING FROM TONGUE (Vascular disorders) | 1
Hemorrhage/Bleeding - Other: BLOOD FROM THE THROAT (Vascular disorders) | 1
Hemorrhage/Bleeding - Other: BLOOD IN COUGH SECRETION (Vascular disorders) | 1
Hemorrhage/Bleeding - Other: BLOOD IN SALIVA (Vascular disorders) | 1
Hemorrhage/Bleeding - Other: BLOOD IN SPUTUM (Vascular disorders) | 1
Hemorrhage/Bleeding - Other: BLOOD TINGLED SALIVA (Vascular disorders) | 1
Hemorrhage/Bleeding - Other: BLOOD TINGLED SPUTUM (Vascular disorders) | 1
Hemorrhage/Bleeding - Other: CATHETER SITE (Vascular disorders) | 1
Hemorrhage/Bleeding - Other: CONJUNCTIVAL RIGHT EYE HEMORRHAGE (Vascular disorders) | 1
Hemorrhage/Bleeding - Other: ECCHYMESIS LEFT AXILLA (Vascular disorders) | 1
Hemorrhage/Bleeding - Other: ECCHYMOSES (Vascular disorders) | 1
Hemorrhage/Bleeding - Other: ECCHYMOSIS AFTER HICKMAN CATHETER REMOVAL (Vascular disorders) | 1
Hemorrhage/Bleeding - Other: GUMS BLEEDING (Vascular disorders) | 1
Hemorrhage/Bleeding - Other: HICKMAN SITE BLEEDING (Vascular disorders) | 1
Hemorrhage/Bleeding - Other: MINIMAL BLEEDING UPON REMOVAL OF HICKMAN CATHETER (Vascular disorders) | 1
Hemorrhage/Bleeding - Other: MOUTH (GUM) BLEEDING (Vascular disorders) | 1
Hemorrhage/Bleeding - Other: MOUTH BLEEDING (Vascular disorders) | 6
Hemorrhage/Bleeding - Other: OOZING OF BLOOD FROM THROAT (Vascular disorders) | 1
Hemorrhage/Bleeding - Other: SCANT AMOUNT OF BLOOD AT HICKMAN CATHETER SITE (Vascular disorders) | 1
Hemorrhage/Bleeding - Other: SCLERAL HEMORRHAGE (Vascular disorders) | 1
Hemorrhage/Bleeding - Other: SLIGHT BLEEDING FROM HICKMAN SITE (Vascular disorders) | 1
Hemorrhage/Bleeding - Other: SLIGHT OOZING FROM BMBX SITE AT PELVIS BONE (Vascular disorders) | 1
Hemorrhage/Bleeding - Other: SUBCONJUNCTIVAL HEMORRHAGE (Vascular disorders) | 1
Hemorrhage/Bleeding - Other: TONGUE BLEEDING (Vascular disorders) | 2
Petechiae/purpura (hemorrhage/bleeding into skin or mucosa) (Vascular disorders) | 6
Hepatobiliary/Pancreas - Other: 2 SOLID LESIONS IN LIVER (Hepatobiliary disorders) | 1
Hepatobiliary/Pancreas - Other: HYPOPROTEINEMIA (Hepatobiliary disorders) | 1
Febrile neutropenia (fever of unknown origin) (Infections and infestations) | 34
Infection - Other: CONTACT ISOLATION DUE TO C. DIFFICILE INFECTION (Infections and infestations) | 1
Infection - Other: SEPSIS (Infections and infestations) | 1
Infection - Other: SPUTUM (MRSA) (Infections and infestations) | 1
Infection - Other: TOXIC SHOCK SYNDROME (Infections and infestations) | 1
Infection - Other: UPPER RESPIRATORY INFECTION (Infections and infestations) | 2
Infection - Other: UTI (MIXED) (Infections and infestations) | 1
Infection with unknown ANC (Infections and infestations) | 11
Infection with grade 3 or 4 neutropenia (Infections and infestations) | 19
Infection with unknown ANC (Infections and infestations) | 4
Infection without neutropenia (Infections and infestations) | 21
Infection, Bacterial (COH) (Infections and infestations) | 24
Infection, Fungal (COH) (Infections and infestations) | 8
Infection, Viral (Infections and infestations) | 17
Lymphatics - Other: SPLENOMEGALY (US) (Blood and lymphatic system disorders) | 1
ALT, SGPT (serum glutamic pyruvic transaminase) (Metabolism and nutrition disorders) | 41
AST, SGOT(serum glutamic oxaloacetic transaminase) (Metabolism and nutrition disorders) | 36
Acidosis (metabolic or respiratory) (Metabolism and nutrition disorders) | 1
Albumin, serum-low (hypoalbuminemia) (Metabolism and nutrition disorders) | 45
Alkaline phosphatase (Metabolism and nutrition disorders) | 27
Alkalosis (metabolic or respiratory) (Metabolism and nutrition disorders) | 2
Bicarbonate, serum-low (Metabolism and nutrition disorders) | 14
Bilirubin (hyperbilirubinemia) (Metabolism and nutrition disorders) | 10
CPK (creatine phosphokinase) (Metabolism and nutrition disorders) | 1
Calcium, serum-high (hypercalcemia) (Metabolism and nutrition disorders) | 3
Calcium, serum-low (hypocalcemia) (Metabolism and nutrition disorders) | 44
Cholesterol, serum-high (hypercholesteremia) (Metabolism and nutrition disorders) | 19
Creatinine (Metabolism and nutrition disorders) | 14
Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 42
Glucose, serum-low (hypoglycemia) (Metabolism and nutrition disorders) | 11
Magnesium, serum-high (hypermagnesemia) (Metabolism and nutrition disorders) | 5
Magnesium, serum-low (hypomagnesemia) (Metabolism and nutrition disorders) | 29
Phosphate, serum-low (hypophosphatemia) (Metabolism and nutrition disorders) | 27
Potassium, serum-high (hyperkalemia) (Metabolism and nutrition disorders) | 3
Potassium, serum-low (hypokalemia) (Metabolism and nutrition disorders) | 40
Sodium, serum-high (hypernatremia) (Metabolism and nutrition disorders) | 7
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 39
Uric acid, serum-high (hyperuricemia) (Metabolism and nutrition disorders) | 8
Muscle weakness, generalized or specific area (not due to neuropathy) (Musculoskeletal and connective tissue disorders) | 5
Musculoskeletal/Soft Tissue - Other: LOWER BACK PAIN (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal/Soft Tissue - Other: SWOLLEN JOINTS OF HANDS (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal/Soft Tissue - Other: SWOLLEN LEFT ELBOW JOINT (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal/Soft Tissue - Other: SWOLLEN LEFT LEG (Musculoskeletal and connective tissue disorders) | 1
Ataxia (incoordination) (Nervous system disorders) | 2
Confusion (Nervous system disorders) | 9
Dizziness (Nervous system disorders) | 20
Extrapyramidal/involuntary movement/restlessness (Nervous system disorders) | 3
Hallucinations (Nervous system disorders) | 5
Mood alteration (Nervous system disorders) | 30
Neurology - Other: ANXIETY (Nervous system disorders) | 1
Neurology - Other: DIURNAL VARIATION OF MOOD (Nervous system disorders) | 1
Neurology - Other: DROWSINESS (Nervous system disorders) | 1
Neurology - Other: FEAR (Nervous system disorders) | 1
Neurology - Other: FEARFUL TO USE FENTANYL BOLUSES (Nervous system disorders) | 1
Neurology - Other: FLAT AFFECT ON PSYCHOSOCIAL ASSESSMENT (Nervous system disorders) | 1
Neurology - Other: FLAT EFFECT (Nervous system disorders) | 1
Neurology - Other: FRUSTRATION (Nervous system disorders) | 1
Neurology - Other: IRRITABILITY (MOOD ALTERATION) (Nervous system disorders) | 1
Neurology - Other: LETHARGY (Nervous system disorders) | 1
Neurology - Other: NERVOUSNESS (Nervous system disorders) | 1
Neurology - Other: NIGHTMARES (Nervous system disorders) | 1
Neurology - Other: NUMBNESS (Nervous system disorders) | 2
Neurology - Other: PANIC ATTACK (Nervous system disorders) | 1
Neurology - Other: RUMINATIVE, OBSESSIVE AND FEARFUL MUCH OF THE TIME (Nervous system disorders) | 1
Neurology - Other: SLEEPINESS (Nervous system disorders) | 2
Neurology - Other: SOMNOLENCE (Nervous system disorders) | 1
Neurology - Other: TINGLING SENSATION (Nervous system disorders) | 1
Neurology - Other: UNSTEADINESS (Nervous system disorders) | 1
Neurology - Other: UNSTEADINESS BECAUSE OF VICODIN (Nervous system disorders) | 1
Neurology - Other: VIBRATING SENSATION AT FEET WHILE WALKING (Nervous system disorders) | 1
Neurology - Other: VIBRATING SENSATION AT TORSO WHILE SITTING (Nervous system disorders) | 1
Neuropathy: cranial (Nervous system disorders) | 1
Neuropathy: motor (Nervous system disorders) | 3
Neuropathy: sensory (Nervous system disorders) | 5
Somnolence/depressed level of consciousness (Nervous system disorders) | 9
Speech impairment (e.g., dysphasia or aphasia) (Nervous system disorders) | 1
Syncope (fainting) (Nervous system disorders) | 2
Tremor (Nervous system disorders) | 4
Dry eye syndrome (Eye disorders) | 8
Nystagmus (Eye disorders) | 2
Ocular surface disease (Eye disorders) | 1
Ocular/Visual - Other: CONGESTED CONJUNCTIVAL (Eye disorders) | 1
Ocular/Visual - Other: CONJUNCTIVITIS (Eye disorders) | 1
Ocular/Visual - Other: DILATATION OF PUPIL (LT. EYE) (Eye disorders) | 1
Ocular/Visual - Other: IRRITATION (Eye disorders) | 1
Ocular/Visual - Other: ITCHINESS OF EYES (Eye disorders) | 1
Ocular/Visual - Other: OD-VITREOUS OPACITY WITHOUT RETINAL DEFECT (Eye disorders) | 1
Ocular/Visual - Other: PERIORBITAL PUFFINESS (Eye disorders) | 1
Ocular/Visual - Other: SLUGGISHNESS AND DILATATION OF RT. EYE PUPIL (Eye disorders) | 1
Ocular/Visual - Other: SWOLLEN EYES (Eye disorders) | 1
Ocular/Visual - Other: TRANSIENT SPOTS IN FRONT OF EYES (Eye disorders) | 1
Ophthalmoplegia/diplopia (double vision) (Eye disorders) | 2
Vision-blurred vision (Eye disorders) | 5
Vision-flashing lights/floaters (Eye disorders) | 2
Watery eye (epiphora, tearing) (Eye disorders) | 2
Pain (General disorders) | 40
Pain - Other: (General disorders) | 1
Pain - Other: ABDOMINAL TENDERNESS (General disorders) | 1
Pain - Other: ACHES AND STRAINS OF CHEST WALL MUSCLES BECAUSE OF COUGHING (General disorders) | 1
Pain - Other: BACK PAIN (General disorders) | 6
Pain - Other: BACK PAIN/BACK SPASM (General disorders) | 1
Pain - Other: BODY ACHES (General disorders) | 2
Pain - Other: BURNING BLOOD-SHOT PAIN EYES (General disorders) | 1
Pain - Other: CATHETER PAIN (General disorders) | 1
Pain - Other: CHEST DISCOMFORT (General disorders) | 1
Pain - Other: CHEST PRESSURE (General disorders) | 1
Pain - Other: CVA TENDERNESS (General disorders) | 1
Pain - Other: DECUBITUS AREA PAIN (General disorders) | 1
Pain - Other: DIFFUSE ACHES AND PAINS (General disorders) | 1
Pain - Other: DIFFUSE BUTTOCK AND SACRAL PAIN DUE TO DECUBITUS ULCER (General disorders) | 1
Pain - Other: EPIGASTRIC PAIN (General disorders) | 1
Pain - Other: EPIGASTRIC PAIN WITH RADIATION TO BACK (General disorders) | 1
Pain - Other: ESOPHAGEAL DISCOMFORT (General disorders) | 1
Pain - Other: ESOPHAGEAL PAIN (General disorders) | 1
Pain - Other: GENERALIZED ACHES AND TENDERNESS (General disorders) | 1
Pain - Other: GENERALIZED BODY ACHES (General disorders) | 1
Pain - Other: HICKMAN CATHETER PAIN (General disorders) | 3
Pain - Other: KNEES PAIN (General disorders) | 1
Pain - Other: LEFT ARM AND SHOULDER PAIN (General disorders) | 1
Pain - Other: LEFT HAND PAIN (General disorders) | 1
Pain - Other: LEFT LEG (General disorders) | 1
Pain - Other: LEG PAIN (General disorders) | 2
Pain - Other: LEGS PAIN (General disorders) | 1
Pain - Other: LOW BACK PAIN WHILE ON RUNNING (General disorders) | 1
Pain - Other: LOWER BACK PAIN (General disorders) | 1
Pain - Other: LT. FLANK PAIN (General disorders) | 1
Pain - Other: LT. KNEE PAIN (General disorders) | 1
Pain - Other: LT. NECK SWELLING (General disorders) | 1
Pain - Other: LT. SHOULDER PAIN (General disorders) | 1
Pain - Other: MOUTH PAIN (General disorders) | 13
Pain - Other: PAIN AT BUTTOCKS DUE TO SHINGLES (General disorders) | 1
Pain - Other: PAIN AT HANDS AND FEET (General disorders) | 1
Pain - Other: PAIN AT HICKMAN CATHETER EXIT SITE (General disorders) | 1
Pain - Other: PAIN AT RAC EXIT SITE (General disorders) | 1
Pain - Other: PAIN AT RUQ (General disorders) | 1
Pain - Other: PAIN DUE TO BP TAKING (General disorders) | 1
Pain - Other: PAIN DUE TO LP PROCEDURE (General disorders) | 1
Pain - Other: PAIN IN PALMS (General disorders) | 1
Pain - Other: PAIN WHILE PASSING BLOOD CLOT IN FOLEY'S CATHETER (General disorders) | 1
Pain - Other: PALM PAIN (General disorders) | 1
Pain - Other: PAROTIDITIS (LT. SIDE) (General disorders) | 1
Pain - Other: RAC SITE DISCOMFORT (General disorders) | 1
Pain - Other: RAC SITE PAIN (General disorders) | 2
Pain - Other: RIGHT ARM SORENESS (General disorders) | 1
Pain - Other: RIGHT FOREARM DISCOMFORT (General disorders) | 1
Pain - Other: RUQ TENDERNESS (General disorders) | 1
Pain - Other: SCROTAL PAIN (General disorders) | 1
Pain - Other: SHOULDER PAIN (General disorders) | 3
Pain - Other: SINUS PAIN (General disorders) | 1
Pain - Other: SORE THROAT (General disorders) | 2
Pain - Other: TENDER PALMS (General disorders) | 1
Pain - Other: TENDERNESS AT H. CATHETER SITE (General disorders) | 1
Pain - Other: TENDERNESS AT HICKMAN CATHETER SITE (General disorders) | 1
Pain - Other: TENDERNESS AT RUQ (General disorders) | 1
Pain - Other: TENDERNESS OVER LEFT CHEECK SWELLING (General disorders) | 1
Pain - Other: TENDERNESS OVER SINUSES (General disorders) | 1
Pain - Other: THROAT PAIN (General disorders) | 16
Pain - Other: TOE AND FINGERTIP PAIN (General disorders) | 1
Pain - Other: TONGUE PAIN (General disorders) | 1
Pain ABDOMINAL CRAMPING (General disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 28
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 11
Hiccoughs (hiccups, singultus) (Respiratory, thoracic and mediastinal disorders) | 7
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 7
Pleural effusion (non-malignant) (Respiratory, thoracic and mediastinal disorders) | 5
Pneumonitis/pulmonary infiltrates (Respiratory, thoracic and mediastinal disorders) | 5
Pulmonary/Upper Respiratory - Other: ASPIRATION PNEUMONIA (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary/Upper Respiratory - Other: ATELECTASIS (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary/Upper Respiratory - Other: ATELECTASIS LLL (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary/Upper Respiratory - Other: ATELECTASIS LT. MID LUNG (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary/Upper Respiratory - Other: ATELECTASIS OF RLL WITH ELEVATED DIAPHRAGM (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary/Upper Respiratory - Other: BIBASILAR RALES (Respiratory, thoracic and mediastinal disorders) | 2
Pulmonary/Upper Respiratory - Other: BILATERAL DIFFUSE RALES (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary/Upper Respiratory - Other: BILATERAL ELEVATION OF HEMIDIAPHRAGM (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary/Upper Respiratory - Other: BILATERAL RHONCHI (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary/Upper Respiratory - Other: BILATERAL SCATTERED CRACKLES (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary/Upper Respiratory - Other: BLUNTING OF LT. COSTOPHRENIC ANGLE (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary/Upper Respiratory - Other: CHEST TIGHTNESS (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary/Upper Respiratory - Other: CHRONIC SNEEZING (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary/Upper Respiratory - Other: CLEAR SPUTUM PRODUCTION (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary/Upper Respiratory - Other: COLD WITH NASAL DISCHARGE (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary/Upper Respiratory - Other: CRACKLES AT LLL LUNGS (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary/Upper Respiratory - Other: CRACKLES AT LUNG BASES (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary/Upper Respiratory - Other: CRACKLES AT RLL (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary/Upper Respiratory - Other: DECREASED BREATH SOUND AT LT. LUNG (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary/Upper Respiratory - Other: DECREASED BREATH SOUND AT LUNG BASES (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary/Upper Respiratory - Other: DECREASED BREATH SOUND RT. LUNG (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary/Upper Respiratory - Other: DECREASED BS AT RLL LUNG (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary/Upper Respiratory - Other: DRY NOSE (Respiratory, thoracic and mediastinal disorders) | 2
Pulmonary/Upper Respiratory - Other: ETHMOID SINUSITIS (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary/Upper Respiratory - Other: EXPIRATORY WHEEZING (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary/Upper Respiratory - Other: MUCUS OBSTRUCTION OF ET TUBE (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary/Upper Respiratory - Other: MUCUS PLUG LLL (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary/Upper Respiratory - Other: NASAL CONGESTION (Respiratory, thoracic and mediastinal disorders) | 4
Pulmonary/Upper Respiratory - Other: NASAL DRAINAGE (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary/Upper Respiratory - Other: NASAL SECRETION (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary/Upper Respiratory - Other: NASAL STUFFINESS (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary/Upper Respiratory - Other: OCCASIONAL RHONCHI (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary/Upper Respiratory - Other: POST-NASAL DRAINAGE (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary/Upper Respiratory - Other: POST-NASAL DRIP (Respiratory, thoracic and mediastinal disorders) | 2
Pulmonary/Upper Respiratory - Other: POSTNASAL DRIP (Respiratory, thoracic and mediastinal disorders) | 2
Pulmonary/Upper Respiratory - Other: PULMONARY EDEMA (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary/Upper Respiratory - Other: PULMONARY VASCULAR CONGESTION (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary/Upper Respiratory - Other: RALES RT. LUNG BASE (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary/Upper Respiratory - Other: RHONCHI BOTH LUNGS (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary/Upper Respiratory - Other: RHONCHI RT. LOWER LOBE (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary/Upper Respiratory - Other: RLL ATELECTASIS (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary/Upper Respiratory - Other: RLL INFILTRATE (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary/Upper Respiratory - Other: RUNNING NOSE (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary/Upper Respiratory - Other: RUNNY NOSE (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary/Upper Respiratory - Other: SINUS CONGESTION (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary/Upper Respiratory - Other: SINUSITIS (Respiratory, thoracic and mediastinal disorders) | 2
Pulmonary/Upper Respiratory - Other: SNEEZING (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary/Upper Respiratory - Other: STUFFY NOSE (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary/Upper Respiratory - Other: SUBSEGMENTAL ATELECTASIS (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary/Upper Respiratory - Other: TACHYPNEA (Respiratory, thoracic and mediastinal disorders) | 2
Pulmonary/Upper Respiratory - Other: UPPER AIRWAY CONGESTION (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary/Upper Respiratory - Other: UPPER AIRWAY SWELLING (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary/Upper Respiratory - Other: WHEEZING (Respiratory, thoracic and mediastinal disorders) | 3
Pulmonary/Upper Respiratory - Other: WHEEZING AFTER BLOOD TRANSFUSION (Respiratory, thoracic and mediastinal disorders) | 1
Voice changes/dysarthria (e.g., hoarseness, loss or alteration in voice, laryngitis) (Respiratory, thoracic and mediastinal disorders) | 18
Bladder spasms (Renal and urinary disorders) | 2
Cystitis (COH) (Renal and urinary disorders) | 1
Incontinence (Renal and urinary disorders) | 1
Renal/Genitourinary - Other: BLOOD CLOT IN FOLEY'S CATHETER (Renal and urinary disorders) | 1
Renal/Genitourinary - Other: BUN ELEVATED (Renal and urinary disorders) | 1
Renal/Genitourinary - Other: DARK ORANGE COLOR URINE (Renal and urinary disorders) | 1
Renal/Genitourinary - Other: DIFFICULTY VOIDING (Renal and urinary disorders) | 1
Renal/Genitourinary - Other: GENITAL SORES (Renal and urinary disorders) | 1
Renal/Genitourinary - Other: INCONTINENCE (Renal and urinary disorders) | 1
Renal/Genitourinary - Other: OBSTRUCTIVE UROPATHY (Renal and urinary disorders) | 1
Renal/Genitourinary - Other: PUL. OTHER/RHONCHI RT. LUNG BASE (Renal and urinary disorders) | 1
Urinary frequency/urgency (Renal and urinary disorders) | 3
Libido (Reproductive system and breast disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2004-04-20): https://cdn.clinicaltrials.gov/large-docs/69/NCT00534469/Prot_SAP_000.pdf